CLINICAL TRIAL: NCT03179956
Title: Biomarker Window of Opportunity Study to Evaluate the Impact of Ribociclib on Head and Neck Squamous Cell Cancer
Brief Title: Impact of Ribociclib on Head and Neck Squamous Cell Cancer
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HN-089
Record Dates: First submitted 2017-06-06; First posted 2017-06-07 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ribociclib (Experimental)
  Interventions: Drug: Ribociclib

INTERVENTIONS:
Drug: Ribociclib — Treatment with ribociclib [600mg] will be from Days 1-14, with surgical resection on Day 14. Labs (CBC, CMP, coagulation parameters) and an ECG will be checked once in a window defined by days 9-12.

SUMMARY:
A window of opportunity study which would allow brief treatment of HPV negative SCCHN with a CDK4/6 inhibitor, in the pre-operative setting, with biomarker analyses of pre and post treatment tissue. Given that the standard treatment for this population is surgical resection, this would not impact or alter standard therapy for this population. The goal will be to learn more about the alterations in pRB1 levels, as well as other signaling markers, in order to be able to eventually plan a biomarker driven treatment study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has an oral cavity cancer, HPV negative oropharynx cancer, or larynx cancer that is amenable to surgical resection for curative intent.
2. Surgical resection must be the part of their standard treatment for management of SCCHN cancer.
3. Patient must have archival tissue and must consent to provide pre-treatment archival tissue.
4. Patient has signed the Informed Consent (ICF) prior to any screening procedures and is able to comply with protocol requirements.
5. Male or Female patients who are 18 years or older.
6. Patients with known central nervous system (CNS) involvement must have clinically stable CNS tumor at the time of screening and should not be receiving steroids and/or enzyme-inducing anti-epileptic medications for brain metastases.
7. Patient has adequate bone marrow and organ function as defined by the following laboratory values at screening:

   * Absolute neutrophil count ≥1.5 × 109/L
   * Platelets ≥100 × 109/L
   * Hemoglobin ≥9.0 g/dL
   * Potassium, total calcium (corrected for serum albumin), magnesium, sodium and phosphorus within normal limits for the institution or corrected to within normal limits with supplements before first dose of study medication per protocol guidelines
   * INR ≤1.5
   * Serum creatinine ≤1.5 mg/dL or creatinine clearance ≥50 mL/min
   * In the absence of liver metastases, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <2.5 x ULN. If the patient has liver metastases, ALT and AST <5 x ULN
   * Total bilirubin < ULN; or total bilirubin ≤3.0 x ULN or direct bilirubin ≤1.5 x ULN in patients with well-documented Gilbert's Syndrome.
8. Standard, triplicate 12-lead ECG with the following parameters (defined as the mean of the triplicate ECGs):

   * QTcF interval at screening <450msec (using Fridericia's correction)
   * Resting heart rate 50-90 bpm
9. Women of child bearing potential must agree to use adequate means to prevent pregnancy
10. Men should either be sterile or must agree not to impregnate a women

Exclusion Criteria:

1. Patients with known hypersensitivity to ribociclib or similar class of agent.
2. Patients with concurrent malignancy which requires active treatment or malignancy within 3 years prior to starting study drug with the exception of basal or squamous cell carcinoma, or non-melanomatous skin cancer.
3. Patients with impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drug (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
4. Patients with known history of HIV infection (testing not mandatory).
5. Patients with any other concurrent severe and/or uncontrolled medical condition that, in the investigator's judgment, would cause unacceptable safety risks, contraindicate patient participation in the clinical study or compromise compliance with the protocol (e.g. chronic pancreatitis, chronic active hepatitis, active untreated or uncontrolled fungal, bacterial or viral infections, etc.).
6. Clinically significant, uncontrolled heart disease and/or recent events including any of the following:

   * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) or symptomatic pericarditis within 12 months prior to screening
   * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
   * Documented cardiomyopathy
   * Patients with Left Ventricular Ejection Fraction (LVEF) <50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO) at screening
   * History of any cardiac arrhythmias, e.g., ventricular, supraventricular, nodal arrhythmias, or conduction abnormality, high grade AV block (e.g. bifascicular block, Mobitz type II and third degree AV block) within 12 months of screening
   * Congenital long QT syndrome or family history of long QT syndrome
   * Risk factors for Torsades de Pointe (TdP) including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia.
   * Concomitant use of medication(s) with a known risk to prolong the QT interval and/or known to cause Torsades de Pointe that cannot be discontinued (within 5 half-lives or 7 days prior to starting study drug) or replaced by safe alternative medication
   * Inability to determine the QT interval on screening (QTcF, using Fridericia's correction)
   * Systolic blood pressure (SBP) >160 mmHg or <90 mmHg at screening
   * Bradycardia (heart rate <50 at rest), by ECG or pulse, at screening
7. Patients receiving any of the following medications that cannot be discontinued 7 days prior to starting study drug (see Appendix II, Table 1 for details):

   1. Known strong inducers or inhibitors of CYP3A4/5, including grapefruit, grapefruit hybrids, pummelos, star-fruit, and Seville oranges
   2. That have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5
   3. That have a known risk to prolong the QT interval or induce Torsades de Pointes, herbal preparations/medications, dietary supplements.
8. Patients receiving or have received systemic corticosteroids ≤ 2 weeks prior to starting study drug or who have not fully recovered from side effects of such treatment. The following uses of corticosteroids are permitted: single doses, topical applications (e.g., for rash), inhaled sprays (e.g., for obstructive airways diseases), eye drops or local injections (e.g., intra-articular).
9. Patients receiving warfarin or other coumadin-derived anticoagulant for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH) or fondaparinux is allowed.
10. Patient who has received radiotherapy ≤4 weeks or limited field radiation for palliation ≤2 weeks prior to starting study drug, and who has not recovered to grade 1 or better from related side effects of such therapy (exceptions include alopecia) and/or in whom ≥25% of the bone marrow (Ellis, 1961) was irradiated.
11. Patient who has had prior treatment for current oral cavity malignancy, except for biopsy for diagnostic purposes.
12. Patient has had major surgery within 14 days prior to starting study drug or has not recovered from major side effects (tumor biopsy is not considered as major surgery).
13. Patient has not recovered from all toxicities due to prior anticancer therapies for a different malignancy to NCI-CTCAE version 4.03 Grade ≤1 (Exception to this criterion: patients with any grade of alopecia and neuropathy grade≤ 2 are allowed to enter the study).
14. Patient with a Child-Pugh score B or C.
15. Patient has a history of non-compliance to medical regimen or inability to grant consent.
16. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Treatment with a CDK4/6 inhibitor, Ribociclib, decreases pRB1 levels in patients with SCCHN of the oral cavity, oropharynx and larynx. | 1-2 months
  pre-treatment to post-treatment changes in pRB1 expression levels will be measured

SECONDARY OUTCOMES:
Change in pre-treatment to post-treatment levels of Ki67 in tissue samples from patients | 2-3 months
Change in pre-treatment to post-treatment levels of ERK1/2 in tissue samples from patients | 2-3 months
Change in pre-treatment to post-treatment levels of phosphorylated-ERK1/2 in tissue samples from patients | 2-3 months
Change in pre-treatment to post-treatment levels of p16 in tissue samples from patients | 2-3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Bauman, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No